CLINICAL TRIAL: NCT03873064
Title: Body Mass Index (BMI) and Quality of Life (QoL) in Cancer Patients
Acronym: BMI-QoL
Status: Recruiting | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Collaborators: S.I.C.O.G. partners (Other)
Responsible Party: Principal Investigator, Vincenzo Formica, Consultant in Medical Oncology, Principal Investigator, University of Rome Tor Vergata
Other Study IDs: R.S. 102.17
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Neoplasm Malignant; Body Weight; Quality of Life
Keywords: BMI; EORTC QLQ-C30; metastatic cancer; localized cancer
MeSH Terms: conditions — Neoplasms; Body Weight; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with solid tumor: All consecutive patients with a histologically confirmed diagnosis of solid tumor referred to any of the Medical Oncology Units of the S.I.C.O.G. cooperative group (http://www.sicog.it/).

SUMMARY:
BMI is a simple and widely recorded variable that may capture obesity or cachexia in cancer patients. How BMI is associated to health-related quality of life (HR-QoL) in such patients is poorly investigated.

High BMI may be associated to obesity, an increased burden of comorbidity, reduced physical activity and, in some settings, to more aggressive oncological disease. On the other hand, low BMI may reflect enhanced weight loss, cachectic syndrome, higher tumor burden and adverse prognostic features which all deteriorate quality of life. The aim of the present study is to evaluate the association of BMI and HR-QoL as measured by the EORTC-QLQ-C30 questionnaire in several cancer settings (such as localized vs metastatic or distinct primary tumors).

DETAILED DESCRIPTION:
Health-related quality of life (HRQoL) might have varied association to body weight in patients with solid cancer[1].

On one hand low body weight may reflect cancer-related anorexia and weight loss and cachectic syndrome which are associated to impaired performance status, deteriorated general conditions and advanced cancer[2]. In such patients the probability of recording a low Body Mass Index (BMI) and concomitantly an inferior Health related quality of life (HRQoL, as patient reported outcome, PRO) is high.

On the other hand, some of the hormonal mediators found at increased concentration in obese patients, such as insulin-like growth factor (IGF), have been demonstrated to be involved in biological pathways that favor an improved HRQoL[3].

Adding further apparent contradiction is the fact that obesity and high BMI may represent in some cancer settings an adverse feature. In particular, obesity is associated with an increased risk of developing certain tumor types and, in some cancer patients with radically resected primary, of cancer relapse[4]. Moreover high BMI carries often an increased burden of comorbidity (e.g. cardiovascular and metabolic diseases)[5] and reduced physical activity. All these factors may reduce HRQoL.

Studies investigating specific associations between BMI and HRQoL in specific cancer settings are therefore warranted.

The present prospective observational cohort study has the aim of investigating the relationship between BMI and PRO-HRQoL as measured by the EORTC-QLQ-C30 questionnaire [6] in different primary tumors (breast, lung, colorectal and others) and in different cancer stages (localized vs metastatic). Patients will be also stratified according to the presence of cardiovascular and metabolic comorbidities, to the Karnofsky Performance status and according to the oncological treatment received (chemotherapy vs radically resected patients on follow-up). If available, retrospective data will be used to train possible predictive models.

STUDY PROCEDURES Study participation will be offered to all consecutive patients with a histologically confirmed diagnosis of solid tumor referred to the Medical Oncology Units of the S.I.C.O.G. cooperative group (http://www.sicog.it/). Upon acceptance, patients will sign an informed consent and be asked to fill out the EORTC QLQ C30 questionnaire.

All common antropometric, demographic, clinical and biochemical variables will be recorded around the moment of first referral (within three months).

Re-assessable variables, including EORTC QLQ-C30 questionnaire re-administration, will be recorded every 4-6 months thereafter. All data will be stored in a prospectively maintained database.

Among recorded data will be: age, sex, weight, height, occupation, civil status, primary tumor site, tumor stage, possible metastatic sites, past and actual type of oncological treatment, pain score, Karnofsky Performance Status, vital signs, routine blood tests Patients will be oncologically managed according to standard practice Association between BMI and EORTC QLQ-C30 will be assesses using regression analyses across the different clinical settings identified.

STATISTICAL CONSIDERATIONS The design of the study hypothesizes that in metastatic patients an improved HR-QoL is associated with high BMI (non-cachectic patients) An 'exact single-stage design' will be followed [7]. According to historical data (endometrial cancer), 50% of patients with BMI < 30 has a high global health status score (GHS) of the EORTC QLQ C30 (i.e. a GHS score ≥ 80%) [8].

The hypothesis to be tested will be H0, P < P0 vs H1, P > P1, where P is the percentage of patients with GHS ≥ 80%. One-tail alpha error of 0.05 and false-negative (beta) rate of 0.2 will be considered. P0 will be set at 50% and P1 at 65%, looking for a 15% increase in the percentage of high GHS score among patients with BMI >30. The H0 hypothesis will be rejected and H1 accepted with a statistical power of 80% if at least 42 patients out of 69 with BMI > 30 will report a GHS score ≥ 80.

Since BMI > 30 is observed in about 10% of all metastatic patients, a total of 690 metastatic patients will be required. Since metastatic patients are about half of all cancer patients referred to Medical Oncology Units, a final sample size of 1380 cancer patients (all stages) will be set as the target number.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of solid tumor
2. Age >18 years
3. Signed informed consent
4. Life expectancy > 12 weeks

Exclusion Criteria:

1. Inability to fill out the EORTC QLQ-C30 questionnaire.
2. Absence of a certain diagnosis of solid tumor (e.g. subjects on screening programs)
3. Diagnosis of second malignancies that might bias results interpretation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with a histologically confirmed diagnosis of solid tumor referred to any of the Medical Oncology Units of the S.I.C.O.G. cooperative group (http://www.sicog.it/).
Sampling Method: Non-Probability Sample
Enrollment: 1380 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2029-01-15 (Estimated); Study Completion 2034-01-15 (Estimated)

PRIMARY OUTCOMES:
relationship between BMI and EORTC-QLQC30 according to tumor stage | Recruitment period of 36 months + follow-up period of 24 months since enrollment of last patient
  To assess the relationship between BMI and EORTC-QLQC30 scores in localized vs metastatic cancer patients

SECONDARY OUTCOMES:
relationship between BMI and EORTC-QLQC30 according to different clinical settings other than stage | Recruitment period of 36 months + follow-up period of 24 months since enrollment of last patient
  - To assess the relationship between BMI and EORTC-QLQC30 scores according to:
  * primary tumor
  * presence vs absence of cardiovascular and/or metabolic comorbidities
  * Performance status
  * Ongoing chemotherapy treatment vs observation in disease-free patients (follow-up)
  * Other clinical and biochemical variables routinely assessed as common practice

CONTACTS AND LOCATIONS:
Overall Officials: Mario Roselli, Study Chair — Tor Vergata University Hospital
Locations (1):
- Tor Vergata University Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lin LL, Brown JC, Segal S, Schmitz KH. Quality of life, body mass index, and physical activity among uterine cancer patients. Int J Gynecol Cancer. 2014 Jul;24(6):1027-32. doi: 10.1097/IGC.0000000000000166. PMID 24927246
- [Background] Martin L, Birdsell L, Macdonald N, Reiman T, Clandinin MT, McCargar LJ, Murphy R, Ghosh S, Sawyer MB, Baracos VE. Cancer cachexia in the age of obesity: skeletal muscle depletion is a powerful prognostic factor, independent of body mass index. J Clin Oncol. 2013 Apr 20;31(12):1539-47. doi: 10.1200/JCO.2012.45.2722. Epub 2013 Mar 25. PMID 23530101
- [Background] Meyerhardt JA, Sloan JA, Sargent DJ, Goldberg RM, Pollak M, Morton RF, Ramanathan RK, Williamson SK, Findlay BP, Fuchs CS. Associations between plasma insulin-like growth factor proteins and C-peptide and quality of life in patients with metastatic colorectal cancer. Cancer Epidemiol Biomarkers Prev. 2005 Jun;14(6):1402-10. doi: 10.1158/1055-9965.EPI-04-0862. PMID 15941948
- [Background] Renehan AG, Tyson M, Egger M, Heller RF, Zwahlen M. Body-mass index and incidence of cancer: a systematic review and meta-analysis of prospective observational studies. Lancet. 2008 Feb 16;371(9612):569-78. doi: 10.1016/S0140-6736(08)60269-X. PMID 18280327
- [Background] Twig G, Yaniv G, Levine H, Leiba A, Goldberger N, Derazne E, Ben-Ami Shor D, Tzur D, Afek A, Shamiss A, Haklai Z, Kark JD. Body-Mass Index in 2.3 Million Adolescents and Cardiovascular Death in Adulthood. N Engl J Med. 2016 Jun 23;374(25):2430-40. doi: 10.1056/NEJMoa1503840. Epub 2016 Apr 13. PMID 27074389
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] A'Hern RP. Sample size tables for exact single-stage phase II designs. Stat Med. 2001 Mar 30;20(6):859-66. doi: 10.1002/sim.721. PMID 11252008
- [Background] Smits A, Lopes A, Das N, Bekkers R, Galaal K. The impact of BMI on quality of life in obese endometrial cancer survivors: does size matter? Gynecol Oncol. 2014 Jan;132(1):137-41. doi: 10.1016/j.ygyno.2013.11.018. Epub 2013 Nov 18. PMID 24262880